CLINICAL TRIAL: NCT04994197
Title: A Study of the Urine Non-invasive Liquid Biopsy in Diagnosis and Recurrence Diagnosis of Urothelial Carcinoma
Brief Title: Urothelial Tumor Risk Genes Detection With Genetron Uro V1 and LC-WGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Hangzhou Genetron Medical Laboratory Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Genetron Uro V1-001
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-06

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: DNA extracted from urine sediment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diagnosis group of patients with urothelial cancer: Patients with painless intermittent gross hematuria during outpatient/emergency/hospitalization diagnose as urothelial carcinoma in this study will be assigned to this group
  Interventions: Other: Observational study only - no intervention
- Diagnosis group of patients with benign urinary diseases: Patients with painless intermittent gross hematuria during outpatient/emergency/hospitalization diagnose as benign urinary diseases in this study will be assigned to this group
  Interventions: Other: Observational study only - no intervention
- Recurrence diagnosis group with urothelial cancer: Patients who were diagnosed with non-muscle invasive urothelial carcinoma and diagnosed as recurrent urothelial carcinoma in this study will be assigned to this group
  Interventions: Other: Observational study only - no intervention
- Recurrence diagnosis group with benign urinary diseases: Patients who were diagnosed with non-muscle invasive urothelial carcinoma and diagnosed as benign urinary diseases in this study will be assigned to this group
  Interventions: Other: Observational study only - no intervention

INTERVENTIONS:
Other: Observational study only - no intervention — Observational study only - no intervention

SUMMARY:
Genetron Uro V1 perform mutation detection of 17 genes and methylation detection of 1 gene by using urine samples and tumor tissue samples. It is a urine liquid biopsy method that has a great supplementary effect on the existing clinical differential diagnosis technology. The main aim of this study is to compare the test results of Genetron Uro V1 with the standard clinical diagnosis results, and analyze the performance of Genetron Uro V1 in the diagnosis and recurrence diagnosis of urothelial carcinoma.

DETAILED DESCRIPTION:
The current diagnosis of urothelial carcinoma is mainly based on imaging examination, urine examination and endoscopy. Imaging examinations include ultrasound, CT, MRI, etc., which have limited clinical value when used alone, and are difficult to meet the demand for qualitative research on tumors. The current common methods are urine exfoliated cytology and fluorescence in situ hybridization (FISH). Urine exfoliative cytology is one of the main methods for diagnosis of urothelial cancer and follow-up after surgery. But the sensitivity of urine exfoliated cytology is about 13%-75%, and the specificity is 85%-100%. FISH can detect chromosomal abnormalities in urine exfoliated cells, and combined with urine exfoliated cytology can greatly improve the sensitivity of diagnosis, but the increased cost of multiple examination methods limits its use in diagnosis and each postoperative follow-up. Endoscopy includes cystoscopy and ureteroscopy. Cystoscopy is the most reliable way to diagnose bladder cancer, and some patients with upper urinary tract urothelial cancer also have bladder cancer. Therefore, cystoscopy is almost the "gold standard" method for the diagnosis of urothelial cancer. For most upper urinary tract urothelial cancers, ureteroscopic biopsy is the only method that can be used to pathological diagnosis before surgical resection. However, endoscopy is an invasive examination, which will cause additional pain and complications to the patient, and the resulting local adhesions or trauma will also increase the risk of postoperative recurrence. The characteristics of urothelial cancer are prone to recurrence. Therefore, there are strict follow-up time and standards after surgery. Endoscopy examination is required every three months or six months, which also increases the pain and expense of patients. Based on the above considerations, finding an accurate, non-destructive and economical urine biopsy diagnosis method is an urgent problem in the clinical research of urothelial cancer. Genetron Uro V1 has sensitivity, specificity, and NPV of the pre-diagnostic test for upper urinary tract urothelial carcinoma reached 92.2%, 91.9%, and 94.1%, respectively. Another urine biopsy method based on low-coverage whole-genome sequencing to detect copy number variation (CNV) in patients with urothelial tumors reported its application performance in the diagnosis of urothelial cancer, and its total sensitivity and specificity reached 80.4% and 94.9%, respectively. This project is to optimize new liquid biopsy methods (Genetron Uro V1 and LC-WGS)that will bring greater benefits to the clinic through more standard and larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis Group：

1. Randomly enrolled hematuria patients in outpatient/emergency/inpatient care
2. Gender is not limited
3. Age ≥18 years old
4. Able to provide 100ml urine sample before cystoscopy
5. At the same time, the following requirements still need to be met:

1) Agree to provide personal basic clinical information, pathology and imaging data for scientific research, and sign scientific research-related informed consent 2) Agree to conduct genetic testing services involved in the trial

Recurrence diagnosis group:

1. A patient diagnosed with non-muscular invasive urothelial carcinoma 2. Follow the guidelines for routine recurrence monitoring standard programs 3. No gender limit 4. Age ≥18 years old 5. All urothelial tumors have been surgically removed 6. Agree to perform cystoscopy and urine exfoliation cytology for each recurrence monitoring 7. At the same time, the following requirements still need to be met:

1. Agree to provide personal basic clinical information, pathology and imaging data for scientific research, and sign scientific research-related informed consent; agree to conduct genetic testing services involved in the trial
2. Agree to conduct genetic testing services involved in the experiment -

Exclusion Criteria:

Diagnosis group:

1. Patients with other non-urothelial malignancies (including prostate cancer and renal cell carcinoma)
2. Patients with secondary urothelial tumors
3. Patients who cannot undergo cystoscopy and urine exfoliative cytology
4. Samples with incomplete pathological information, and samples with positive case information that cannot clarify the pathological results and tumor staging
5. Contaminated samples
6. Patients whose urine samples fail to pass the quality control due to reasonable reasons and cannot be sampled again
7. Samples that cannot be tested due to reasonable reasons
8. The researcher believes that there are any conditions that may harm the subject or cause the subject to fail to meet or perform the research requirements
9. Patients who cannot provide written informed consent

Recurrence diagnosis group:

1. Patients with other non-urothelial malignancies (including prostate cancer and renal cell carcinoma)
2. Patients who cannot undergo cystoscopy and urine exfoliative cytology
3. Patients planning to undergo cystectomy/neoadjuvant chemotherapy/radiotherapy
4. Patients who have been enrolled at the pre-recurrence monitoring time point
5. Samples with incomplete pathological information, samples for which the information of positive cases cannot clarify the pathological results and tumor staging
6. Contaminated samples
7. Patients whose urine samples fail to pass the quality control due to reasonable reasons and cannot be sampled again
8. Samples that cannot be tested due to reasonable reasons
9. The researcher believes that there are any conditions that may harm the subject or cause the subject to fail to meet or perform the research requirements
10. Patients who cannot provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with painless intermittent gross hematuria in outpatient/emergency/hospitalization;
  Patients diagnosed with non-muscular invasive urothelial carcinoma;
Sampling Method: Probability Sample
Enrollment: 970 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 18 month
  The sensitivity of Genetron Uro V1 and LC-WGS in the auxiliary diagnosis and recurrence diagnosis of urothelial carcinoma
Specificity | 18 month
  The specificity of Genetron Uro V1 and LC-WGS in the auxiliary diagnosis and recurrence diagnosis of urothelial carcinoma
Positive predictive value (PPV) | 18 month
  The positive predictive value (PPV) of Genetron Uro V1 and LC-WGS in the auxiliary diagnosis and recurrence diagnosis of urothelial carcinoma
Negative predictive value (NPV) | 18 month
  The negative predictive value (NPV) of Genetron Uro V1 and LC-WGS in the auxiliary diagnosis and recurrence diagnosis of urothelial carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Danfeng Xu, Principal Investigator — Ruijin Hospital; Yiming Liang, Study Director — Hangzhou Genetron Medical Laboratory Co., Ltd.
Locations (9):
- China (9):
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Nanjing Zhongda Hospital, Nanjing
  - Luwan Branch of Shanghai Ruijin Hospital, Shanghai
  - Shanghai Fourth People's Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Wuxi People's Hospital, Wuxi
  - Xuzhou Central Hospital, Xuzhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu Y, Ma X, Ai X, Gao J, Liang Y, Zhang Q, Ma T, Mao K, Zheng Q, Wang S, Jiao Y, Zhang X, Li H. A Urine-Based Liquid Biopsy Method for Detection of Upper Tract Urinary Carcinoma. Front Oncol. 2021 Feb 9;10:597486. doi: 10.3389/fonc.2020.597486. eCollection 2020. PMID 33634022
- [Derived] Huang H, Liu A, Liang Y, Xin Y, Liu J, Hao Y, Huang D, Chen L, Li W, Jiang G, Huang Y, Xu Y, Zhang J, Ma T, Xu D, Gao Y. A urinary assay for mutation and methylation biomarkers in the diagnosis and recurrence prediction of non-muscle invasive bladder cancer patients. BMC Med. 2023 Sep 19;21(1):357. doi: 10.1186/s12916-023-03065-5. PMID 37726806
- See also: The diagnostic performance of Gentron Uro V1 in the upper urinary tract urothelial carcinoma — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7901537/